CLINICAL TRIAL: NCT04984421
Title: IMplementation and Evaluation of the School-based Family Support PRogramme A Healthy School Start to Promote Child Health and Prevent OVErweight and Obesity (IMPROVE) - Study Protocol for a Cluster-randomized Trial
Brief Title: IMplementation of the Family Support PRogramme A Healthy School Start to Prevent OVErweight and Obesity (IMPROVE)
Acronym: IMPROVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Liselotte Schäfer Elinder, professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2020-01198
Record Dates: First submitted 2021-07-12; First posted 2021-07-30 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Pediatric Obesity; Overnutrition, Child; Prediabetic State; Diabetes Mellitus, Type 2; Overweight, Childhood
Keywords: BMI; Fidelity; Hybrid type 3 design; Health promotion; Implementation strategies; Primary health care; School health care; Nutrition
MeSH Terms: conditions — Pediatric Obesity; Child Nutrition Disorders; Prediabetic State; Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Cluster randomized controlled trial with a hybrid type 3 evaluation design
Who Masked: Participant
Masking Description: Researchers and school personnel will not be blinded to group allocation, but parents and children will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Basic (Active Comparator): All schools will receive the HSS program. Schools randomly assigned to group 1 will receive implementation strategy bundle 1 (Basic).
  Interventions: Behavioral: Healthy School Start
- Enhanced (Experimental): All schools will receive the HSS program. Schools randomly assigned to group 2 will receive implementation strategy bundle 1+2 (Enhanced).
  Interventions: Behavioral: Healthy School Start

INTERVENTIONS:
Behavioral: Healthy School Start — The Healthy School Start program is a universal 4-component family support program for children starting school (5-7 years of age) promoting healthy dietary habits and physical activity in the home environment to prevent childhood obesity and parents' risk of developing type 2 diabetes. It is targeting both children and parents.

SUMMARY:
IMPROVE is an implementation study aiming to explore the effects of two bundled implementation strategies on the intervention fidelity of the Healthy School Start program (primary outcome) while simultaneously monitoring effects on health outcomes of children and parents (secondary outcomes). Thirty schools in two municipalities will receive the HSS program reaching about 1400 families per school year, for two years.

DETAILED DESCRIPTION:
IMPROVE aims to conduct a hybrid type 3 evaluation design to test the effects of bundled implementation strategies on the intervention fidelity (primary outcome) of the Healthy School Start (HSS) program while simultaneously monitoring effects on health outcomes of children and parents (secondary outcomes). The HSS is a 4-component family support program for children starting school (5-7 years of age) promoting healthy dietary habits and physical activity in the home environment to prevent childhood obesity and parent risk of developing type 2 diabetes.

IMPROVE is a cluster-randomized controlled trial with two arms to evaluate and compare the effects of two different bundles of implementation strategies on intervention fidelity expressed as adherence and responsiveness at 12 and 24 months. Thirty schools in two municipalities will participate in the study reaching about 1400 families per school year. In stakeholder workshops, key implementation determinants were identified according to the domains of the Consolidated Framework for Implementation Research. Through a consensus process with stakeholders, two bundles of implementation strategies were tailored to address context-specific determinants. Schools randomly assigned to group 1 will receive bundle 1 (Basic) and group 2 will receive bundle 1+2 (Enhanced), consisting mainly of external facilitation, fidelity monitoring and feedback strategies. Secondary outcomes will include acceptability, appropriateness, feasibility, organisational readiness as perceived by school staff, child weight status and diet, and parents' risk of type 2 diabetes. Linear and ordinal regression analysis will be used to test the effect on the primary and secondary outcomes, taking clustering into consideration where needed. Process evaluation will be conducted through key stakeholder interviews to investigate experiences of the program and stakeholder perceptions on sustainability.

This systematic approach to investigating the effects of two different bundles of implementation strategies tailored to context-specific determinants on the fidelity of the HSS intervention will provide new insight into feasible implementation strategies and the external supports needed for a school-based health program like the HSS to be effective and sustainable. Results will help inform how to bridge the gap between the research on school-based health programs and routine practice in schools.

ELIGIBILITY:
Inclusion Criteria:

* All children and their parents at the included schools. All involved personnel at the included schools

Exclusion Criteria:

* No

Ages: 5 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1634 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Change in fidelity (A) assessed by questionnaire to parents and school staff | Measured at 12 and 24 months
  Adherence to the four HSS components by indicators developed for this study. Information will be gathered through attendance logs and questionnaires to school staff and parents.
Change in fidelity (R) assessed by questionnaire to parents | Measured at 12 and 24 months
  Responsiveness to the four HSS components by indicators developed for this study. Information will be gathered through questionnaires to parents.

SECONDARY OUTCOMES:
Change in acceptability of the HSS program assessed by questionnaire | Measured at baseline, 12, 24, and 36 months
  Feasibility of implementing the intervention as perceived by school staff, measured with the questionnaire developed by Weiner et al.
Change in appropriateness of the HSS program measured by questionnaire | Measured at baseline, 12, 24, and 36 months
  Appropriateness of implementing the intervention as perceived by school staff, measured with the questionnaire developed by Weiner et al.
Change in feasibility of the HSS program measured by questionnaire | Measured at baseline, 12, 24, and 36 months
  Feasibility of implementing the intervention as perceived by school staff, measured with the questionnaire developed by Weiner et al.
Change in Organisational readiness of school principals assessed by questionnaire | Measured at baseline, 12, 24, and 36 months
  Organisational readiness to change as perceived by school principals with the Leader Readiness to Implement Tool (LRIT)
Change in Organisational readiness by school staff assessed by questionnaire | Measured at baseline, 12, 24, and 36 months
  Organisational readiness to change as perceived by school nurses and teachers with the Staff Readiness to Implement Tool (SRIT)
Fidelity to implementation strategies assessed by checklist | May each year
  Assessment based on checklist developed for this study. Each strategy will be graded as 0=not implemented, 1=partially implemented, 2=fully implemented.
Change in child weight status assessed through measurement of height (m) and weight (kg) | Measured at baseline and after 24 months
  Child BMI will be calculated as in kg/m^2. Weight status will be assessed using age-appropriate BMI cut-off values for thinness, overweight and obesity according to the International Obesity Task Force.
Change in child BMI z-score assessed through measurement of height (m) and weight (kg) | Measured at baseline and after 24 months
  Child BMI will be calculated as in kg/m^2. The BMI z-score will be calculated according to a Swedish reference standard (Karlberg).
Change in child diet assessed by parent questionnaire | Baseline, 12 months, and 24 months
  Dietary indicator foods (fruit, vegetables and energy-dense products) assessed by the diet portion of the Eating and Physical Activity Questionnaire (EPAQ)
Change in parental feeding practices assessed by parent questionnaire | Baseline, 12 months, and 24 months
  Assessed with the Swedish short version of the Comprehensive Feeding Practices Questionnire (CFPQ)
Change in parents' risk of type 2 diabetes assessed by FINDRISC questionnaire | Measured at Baseline, 12 months, and 24 months
  The FINDRISC self-evaluation test to calculate risk of developing type 2 diabetes on a scale from 0-26 points

CONTACTS AND LOCATIONS:
Overall Officials: Liselotte S Elinder, PhD, Principal Investigator — Karolinska Institutet
Locations (3):
- Sweden (3):
  - Municipality, Huddinge, Stockholm County
  - Municipality, Sigtuna, Stockholm County
  - Municipality, Södertälje, Stockholm County

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Annerstedt KS, Ahlgren JA, Patterson E, Andermo S, Norman A, Raposo S, Kwak L, Elinder LS. Comparing tailored implementation strategies to improve intervention fidelity in a school-based obesity prevention program: the IMPROVE hybrid type III trial. Implement Sci. 2025 Dec 28. doi: 10.1186/s13012-025-01481-0. Online ahead of print. PMID 41455974
- [Derived] Elinder LS, Wiklund CA, Norman A, Stattin NS, Andermo S, Patterson E, Hemmingsson E, Cook C, Raposo S, Kwak L. IMplementation and evaluation of the school-based family support PRogram a Healthy School Start to promote child health and prevent OVErweight and obesity (IMPROVE) - study protocol for a cluster-randomized trial. BMC Public Health. 2021 Sep 6;21(1):1630. doi: 10.1186/s12889-021-11663-2. PMID 34488691
- See also: Project website — https://ki.se/gph/en-frisk-skolstart